CLINICAL TRIAL: NCT06211842
Title: Genetic Variations That Increase the Risk for Calcium Kidney Stones: a Family-based Study
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM PAT0295
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Urolithiasis
Keywords: gene polymorphisms
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from stored whole blood will be retained for use in other studies subject to the consent of the participants (46 consented). DNA from 1 participant who did not consent to this will be discarded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many things, like not drinking enough fluids, contribute to making kidney stones and there is also a genetic tendency. We looked into this in 1998-2000 in 14 families with several stone-formers. In four of these the risk for stones was passed down through one line of the family. We have now had a close look at the DNA of 47 members of these four families using a very sensitive technique called exome sequencing. We wanted to see if these individuals had inherited any rare changes (variations) in their DNA which would add to their risk of making stones. We found 11 variations which might be important. Surprisingly, these were not in genes which have been regarded as the main causes of stones. Most of them are unfamiliar to clinicians and scientists world-wide. Experts on the genes gave us helpful advice about the likely significance of the variations. Researchers in Paris, Lille and the UK (Oxford, Cambridge and Sheffield) did analyses to help to decide this. An exciting finding was that one of the variants, not previously identified in stone formers, had just been found in a large Italian family with stones. This small study has shown that: variations in a wide range of genes may contribute to stone formation; these occur in genes that we have not come across before; further laboratory studies are essential to investigate potentially important variants; sharing findings between laboratories doing similar studies world-wide is crucial.

DETAILED DESCRIPTION:
Background:

There is an underlying genetic component to formation of calcium kidney stones, with heritability estimated at about 50%. In most stone formers, genetic susceptibility is polygenic with co-inheritance of multiple small effect gene variants. Genome wide association studies have identified common polymorphisms in 31 genes associated with stone formation. Like other complex polygenic disorders, these do not fully account for genetic susceptibility. Rare/low-frequency variants are also likely to contribute.

In this small observational study, DNA was analysed from members of four calcium stone-forming families in which the risk for stones showed apparent autosomal dominant inheritance. The findings were related to biochemical data obtained in earlier investigations.

Primary objective: to identify rare gene variants associated with stone formation.

Secondary aim: to look for association of the variants with biochemical risk factors for stones recorded in 1998-2000.

Study participants In 1998 to 2000, fourteen families with at least three first-degree relatives who produced calcium stones participated in a study to look for segregation of five genes associated with stone formation. They had biochemical investigations and DNA was analysed using microsatellites. The results were negative. In four of the families, stones had apparent autosomal domain inheritance. Forty- seven of their members were recruited to the new study.

Methods DNA extracted from stored frozen blood was analysed by whole exome sequencing (WES) from ten stone formers (three from each of three families and one from the fourth), and from three members from one kindred who had low excretion of urinary citrate, a stone risk factor. Sequence data were first cross-referenced against a panel of 367 candidate genes reported to be associated with stones, intermediate traits and renal function. Since nephrolithiasis is a relatively common condition, a minor allele frequency of less than or equal to 2% (MAF≤0.02) was applied to retain rare and low frequency variants. We then analysed all other variants from across the genome that were present in all three stone formers within each family that underwent WES. We applied aggressive filtering to this very large dataset. The relevance of each variant to stones was reviewed using the DISEASE database and extensive literature review, and those considered to be significant were prioritised. To examine the association of variants selected for each kindred with stones, they were tracked across the pedigree by Kaspar analysis of DNA from all family participants. [1] Results summary

1 Collectively 20 rare variants (polymorphisms) predicted in silico to be pathogenic and potentially relevant to urolithiasis were identified in the stone formers. Tracking studies for 9 variants showed poor segregation with stones arguing against (but not excluding) a role in stone formation.

2. The clutch of variants was different for each family. 3. Surprisingly, the variants were not in genes which have been regarded as the main causes of stones. Most of them are unfamiliar to clinicians and scientists world-wide.

4. To assess the likely significance of our prioritised variants, we obtained advice from the few groups world-wide with a research interest in the relevant genes. Researchers in Paris, Lille and the UK (Oxford, Cambridge and Sheffield) did preliminary functional analyses to help. However, none had the capacity to do more.

5. From the exome sequences one variant was reported as a pathogenic variant of TCAF2*, the gene for a protein that inactivates a plasma membrane calcium channel. This variant was ultimately demonstrated to be in an inactive pseudogene and not significant.

6 At the time of our study one variant, in the mitochondrial Mg-ATP transporter SLC25A25*, not previously identified in stone formers, was found in a large Italian family with stones. [1] 7. Stone formers with the SLC25A25 and MEPE* variants had phosphaturia. 8. No rare variants associated with low citrate excretion in the family investigated.

Conclusions i) Variations in a wide range of genes may contribute to stone formation; these occur in genes that we have not come across before. ii) Further laboratory studies are essential to investigate potentially important variants, but this is seldom achievable because of limited capacity world-wide to investigate the genes involved. iii) Results reported from exome screens are fallible - pseudogenes are one source of error. iv) Sharing findings between laboratories doing similar studies world-wide is crucial.

* TCAF2 TRPM8 Channel-Associated Factor 2; SLC25A25 Solute Carrier Family 25 Member 25; MEPE matrix extracellular phosphoglycoprotein.

[1] Jabalameli MR, Fitzpatrick FM , Colombo R et al. Exome sequencing identifies a disease variant of the mitochondrial ATP-Mg/Pi carrier SLC25A25 in two families with kidney stones Mol Genet Genomic Med. 2021 Dec;9(12):e1749. doi: 10.1002/mgg3.1749.

ELIGIBILITY:
Inclusion Criteria:

* Stone-forming families who participated in our 1998-2000 study
* Apparent autosomal dominant inheritance of stones transmitted through one line of the family.
* Calcium kidney stone formers.
* Men and women aged 18 year or over.

Exclusion criteria.

* A known hereditary cause of stones
* Children under 18 years of age.
* Uric acid stone formers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four families met the above criteria. A total of 77 family members in primary care were eligible. Of these: 71 were contacted: 47 were recruited; 3 declined; and 21 did not respond to two letters of invitation
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Gene variants linked to kidney stone formation | up to 12 months from end of the study to complete functional studies of identified variants
  The number of stone-formers within a kindred with a gene variant relevant to stones compared with the number of non-stone formers with the variant in the kindred. Stone formation ascertained from interviews with family members in 1998-2000, follow-up questionnaires in 2016 and hospital records.

SECONDARY OUTCOMES:
Gene variants linked to biochemical traits which increase the risk for kidney stones. | up to 12 months from end of the study to complete functional studies of identified variants
  All participants were tested in 1998-2000 for fifteen well recognised biochemical abnormalities which increase stone risk. For each risk factor, pedigree members are now categorised as to whether they had the biochemical abnormality or not. For those with the abnormality, the number with an abnormal gene variant are compared with the number without. Similarly for those with normal biochemical values, the number with a gene variant and the number without are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cook, MRCPPhDFRCPa, Principal Investigator — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient data will be shared with a responsible investigator through a personal request to Dr Valerie Walker or the PI
Supporting Information: Study Protocol, ICF
Time Frame: When the request for information is made & has been approved by Dr Walker or the PI. No time limit since this is anonymised data
Access Criteria: Email approach to Dr Walker or the PI who will review the request. Details of the gene variants found and biochemical data from the original study will be shared.

REFERENCES:
- [Background] Jabalameli MR, Fitzpatrick FM, Colombo R, Howles SA, Leggatt G, Walker V, Wiberg A, Kunji ERS, Ennis S. Exome sequencing identifies a disease variant of the mitochondrial ATP-Mg/Pi carrier SLC25A25 in two families with kidney stones. Mol Genet Genomic Med. 2021 Dec;9(12):e1749. doi: 10.1002/mgg3.1749. Epub 2021 Aug 4. PMID 34346195